CLINICAL TRIAL: NCT03397264
Title: Phase 1b/2a Study of OPT-302 in Combination With Aflibercept for Persistent Central-involved Diabetic Macular Edema
Brief Title: A Dose Ranging Study of OPT-302 With Aflibercept for Persistent Diabetic Macular Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opthea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-302-1003
Record Dates: First submitted 2018-01-01; First posted 2018-01-11 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Phase 1b - sequential dose followed by Phase 2a - parallel arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ph 1b open label; Ph 2a quadruple masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ph 1b: 2.0 mg aflibercept with 0.3 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection (0.05 mL) followed by 0.3 mg OPT-302 intravitreal injection (0.05 mL)
  Interventions: Biological: Aflibercept; Biological: OPT-302
- Ph 1b: 2.0 mg aflibercept with 1.0 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection (0.05 mL) followed by 1.0 mg OPT-302 intravitreal injection (0.05 mL)
  Interventions: Biological: Aflibercept; Biological: OPT-302
- Ph 1b: 2.0 mg aflibercept with 2.0 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection (0.05 mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05 mL)
  Interventions: Biological: Aflibercept; Biological: OPT-302
- Ph 2a: 2.0 mg aflibercept with 2.0 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection (0.05 mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05 mL)
  Interventions: Biological: Aflibercept; Biological: OPT-302
- Ph 2a: 2.0 mg aflibercept with sham (Sham Comparator): 2.0 mg aflibercept intravitreal injection (0.05 mL) followed by sham intravitreal injection
  Interventions: Biological: Aflibercept; Other: Sham intravitreal injection

INTERVENTIONS:
Biological: Aflibercept — Intravitreal injection
  Other Names: Eylea
Biological: OPT-302 — Intravitreal Injection
  Arms: Ph 1b: 2.0 mg aflibercept with 0.3 mg OPT-302; Ph 1b: 2.0 mg aflibercept with 1.0 mg OPT-302; Ph 1b: 2.0 mg aflibercept with 2.0 mg OPT-302; Ph 2a: 2.0 mg aflibercept with 2.0 mg OPT-302
Other: Sham intravitreal injection — Sham (mock) intravitreal injection
  Arms: Ph 2a: 2.0 mg aflibercept with sham

SUMMARY:
A two part, multi-center study consisting of a Phase 1b open label, sequential dose escalation followed by a Phase 2a randomized, double-masked, dose expansion evaluating OPT-302 in combination with aflibercept in participants with persistent central-involved Diabetic Macular Edema.

DETAILED DESCRIPTION:
Study OPT-302-1003 was designed as a 2-part, multicenter study consisting of a Phase 1b open-label, sequential dose escalation followed by a Phase 2a randomized, parallel-group, sham-controlled, double-masked, dose-expansion evaluating intravitreal OPT-302 in combination with aflibercept in participants with persistent central-involved diabetic macula edema.

ELIGIBILITY:
Inclusion Criteria:

* History of diabetic macular edema (DME) ≤ 2 year
* Persistent DME despite prior intravitreal anti-VEGF-A therapy with a sub-optimal response
* Three or more prior anti-VEGF-A therapy intravitreal injections
* EDTRS BCVA score ≤ 73 and ≥ 24 letters

Exclusion Criteria:

* Ocular disorders or ocular treatments which may interfere with assessment of visual acuity, assessment of toxicity, or fundus photography in the Study Eye
* HbA1c ≥ 12% and/or recent signs of uncontrolled diabetes
* Any clinically significant disorder or condition or disease (e.g. cardiovascular, renal conditions) that would make the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Opthea, Study Director — Opthea Limited
Locations (48):
- United States (34):
  - Opthea Investigational Site, Phoenix, Arizona
  - Opthea Investigational Site, Bakersfield, California
  - Opthea Investigational Site, Beverly Hills, California
  - Opthea Investigational Site, Redlands, California
  - Opthea Investigational Site, Sacramento, California
  - Opthea Investigational Site, Santa Ana, California
  - Opthea Investigational Site, Colorado Springs, Colorado
  - Opthea Investigational Site, Boynton Beach, Florida
  - Opthea Investigational Site, Fort Myers, Florida
  - Opthea Investigational Site, Melbourne, Florida
  - Opthea Investigational Site, Pensacola, Florida
  - Opthea Investigational Site, St. Petersburg, Florida
  - Opthea Investigational Site, Augusta, Georgia
  - Opthea Investigational Site, Indianapolis, Indiana
  - Opthea Investigational Site, Des Moines, Iowa
  - Opthea Investigational Site, Wichita, Kansas
  - Opthea Investigational Site, Hagerstown, Maryland
  - Opthea Investigational Site, Las Vegas, Nevada
  - Opthea Investigational Site, Reno, Nevada
  - Opthea Investigational Site, Asheville, North Carolina
  - Opthea Investigational Site, Charlotte, North Carolina
  - Opthea Investigational Site, Youngstown, Ohio
  - Opthea Investigational Site, Portland, Oregon
  - Opthea Investigational Site, Charleston, South Carolina
  - Opthea Investigational Site, West Columbia, South Carolina
  - Opthea Investigational Site, Rapid City, South Dakota
  - Opthea Investigational Site, Germantown, Tennessee
  - Opthea Investigational Site, Abilene, Texas
  - Opthea Investigational Site, Arlington, Texas
  - Opthea Investigational Site, Austin, Texas
  - Opthea Investigational Site, Houston, Texas
  - Opthea Investigational Site, McAllen, Texas
  - Opthea Investigational Site, San Antonio, Texas
  - Opthea Investigational Site, Willow Park, Texas
- Australia (4):
  - Opthea Investigational Site, Parramatta, New South Wales
  - Opthea Investigational Site, Sydney, New South Wales
  - Opthea Investigational Site, Westmead, New South Wales
  - Opthea Investigational Site, Perth, Western Australia
- Israel (8):
  - Opthea Investigational Site, Be’er Ya‘aqov
  - Opthea Investigational Site, Haifa
  - Opthea Investigational Site, Jerusalem
  - Opthea Investigational Site, Kfar Saba
  - Opthea Investigational Site, Petah Tikva
  - Opthea Investigational Site, Rehovot
  - Opthea Investigational Site, Tel Aviv
  - Opthea Investigational Site, Tiberias
- Latvia (2):
  - Opthea Investigational Site, Jelgava
  - Opthea Investigational Site, Riga

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham
Started | 3 | 3 | 3 | 96 | 48
Completed (Completed the Treatment Phase to Week 12) | 3 | 3 | 3 | 89 | 47
Not Completed | 0 | 0 | 0 | 7 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham | Total
Number analyzed (Participants) | 3 | 3 | 3 | 96 | 48 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 58 | 32 | 96
  >=65 years | 1 | 2 | 0 | 38 | 16 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Ph1b and Ph2a studies were two separate studies within the one protocol. Combined mean age across the two studies was not calculated.
  years
    Ph 1b: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 9
    Ph 1b | 59.0 (6.24) | 68.7 (7.51) | 55.7 (7.02) |  |  | 61.1 (8.39)
    Ph 2a: number analyzed (Participants) | 0 | 0 | 0 | 96 | 48 | 144
    Ph 2a |  |  |  | 61.8 (10.07) | 61.2 (9.40) | 61.6 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 36 | 18 | 56
  Male | 2 | 2 | 3 | 60 | 30 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 8 | 8 | 17
  White | 3 | 2 | 3 | 87 | 37 | 132
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Latvia | 0 | 0 | 0 | 6 | 3 | 9
  United States | 3 | 3 | 3 | 61 | 31 | 92
  Israel | 0 | 0 | 0 | 24 | 10 | 34
  Australia | 0 | 0 | 0 | 5 | 4 | 9
Baseline ETDRS Best Corrected Visual Acuity [Mean (Standard Deviation); unit: Letters read] | 64.3 (7.02) | 64.7 (1.53) | 66.0 (8.89) | 63.3 (8.31) | 63.9 (9.44) | 63.5 (8.68)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Safety and Tolerability will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events and CTC v4.0 (if available, otherwise protocol defined grading were used)
Time Frame: Baseline to Week 12
Population: Safety Population; Ph2a: One participant assigned 2.0 mg OPT-302 with aflibercept did not receive OPT-302 therefore this participant was analyzed as part of the sham combination for the safety analysis only.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 3 | 3 | 3 | 95 | 49
Participants
  Treatment Emergent AE to Wk 12 | 3 | 2 | 1 | 59 | 28
  Ocular Treatment Emergent AEs to Wk 12 | 2 | 2 | 1 | 43 | 16
  Non-ocular Treatment Emergnt AEs to Wk 12 | 2 | 2 | 0 | 35 | 17
  Ocular SAEs to Wk 12 | 0 | 0 | 0 | 0 | 0
  Non Ocular SAEs to Wk 12 | 1 | 1 | 0 | 8 | 1

2. Primary Outcome: Phase 2a: Response Rate Defined as Proportion of Participants Receiving OPT-302 With Aflibercept Achieving at Least a 5-letter Gain in BCVA at Week 12
Description: Change from baseline in Best Corrected Visual Acuity (BCVA) will be measured at Week 12 according to Early Treatment Diabetic Retinopathy Score (ETDRS) criteria
Time Frame: Baseline to Week 12
Population: Primary Analysis (pre-specified) OPT-302 combination therapy will be considered to have clinical activity if >= 27 of 72 participants have a >= 5 letters gain in BCVA from baseline to week 12. The combination therapy will be considered to have insufficient clinical activity if <= 25 of 72 participants have a >= 5 letters gain in BCVA from baseline to week 12.
Measure: Count of Participants; unit: Participants
Groups:
- Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05 mL) followed highest tested or maximum tolerated dose from Phase 1b OPT-302 intravitreal injection (0.05 mL) (2.0 mg)
  Aflibercept: Intravitreal injection
  OPT-302: Intravitreal Injection
Arm/Group | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302
Number analyzed (Participants) | 72
Participants | 38

3. Secondary Outcome: Mean Change in BCVA
Description: Mean change in Best Corrected Visual Acuity (BCVA). BCVA will be measured according to Early Treatment Diabetic Retinopathy Score (ETDRS) criteria
Time Frame: Baseline to Week 12
Population: Per Protocol Population
Measure: Mean (Standard Error); unit: Letters
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 3 | 3 | 3 | 75 | 40
Letters | 3.0 (2.52) | 5.7 (1.20) | 14.3 (5.46) | 5.9 (0.79) | 6.1 (0.96)

4. Secondary Outcome: Mean Change in CST
Description: Mean change in central subfield thickness (CST) on spectral domain coherence tomography (SD-OCT)
Time Frame: Baseline to Week 12
Population: Per Protocol Population; and where CST measurements at Week 12 were available to assess the endpoint.
Measure: Mean (Standard Error); unit: µm
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 3 | 3 | 3 | 74 | 39
µm | -116.0 (46.12) | -41.0 (28.88) | -57.0 (12.86) | -52.2 (10.28) | -34.9 (12.01)

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: Ph2a: One participant assigned 2.0 mg OPT-302 with aflibercept did not receive OPT-302 therefore this participant was analysed as part of the sham combination for the safety analysis only.
Arm/Group | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 | Ph 2a: 2.0 mg Aflibercept With Sham
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/95 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 8/95 | 1/49
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 36/95 | 15/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 (N=3) | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 (N=3) | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 (N=3) | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 (N=95) | Ph 2a: 2.0 mg Aflibercept With Sham (N=49)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ocular SAE (Eye disorders) | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph 1b: 2.0 mg Aflibercept With 0.3 mg OPT-302 (N=3) | Ph 1b: 2.0 mg Aflibercept With 1.0 mg OPT-302 (N=3) | Ph 1b: 2.0 mg Aflibercept With 2.0 mg OPT-302 (N=3) | Ph 2a: 2.0 mg Aflibercept With 2.0 mg OPT-302 (N=95) | Ph 2a: 2.0 mg Aflibercept With Sham (N=49)
Conjunctival Haemorrhage (Eye disorders) | 1 | 1 | 1 | 19 | 6
Intraocular Pressure Increased (Eye disorders) | 0 | 0 | 0 | 13 | 3
Punctate Keratitis (Eye disorders) | 1 | 0 | 0 | 2 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator may publish data or results from the Study; provided the Principal Investigator submits the proposed publication to Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary and/or commercially sensitive to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT03397264/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03397264/SAP_001.pdf